CLINICAL TRIAL: NCT03519126
Title: Efficacy of Vaginal and Transcutaneous Electrostimulation of the Posterior Tibial Nerve in the Treatment of Overactive Bladder
Brief Title: Electrostimulation in the Treatment of Idiopathic Overactive Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the covid-19 pandemic
Sponsor: Janaina Mayer de Oliveira Nunes (Other)
Responsible Party: Sponsor-Investigator, Janaina Mayer de Oliveira Nunes, Master, Universidade Federal do Piauí
Organization: Universidade Federal do Piauí (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Overactive bladder
Record Dates: First submitted 2018-04-12; First posted 2018-05-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urinary Bladder, Overactive; Electric Stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: It is a randomized, controlled, simple blind trial with comparative analysis between study groups and a control, performed in three moments: pre and post clinical intervention and one month after the end of treatment (follow up).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vaginal (Experimental): Group of volunteers who will be treated with vaginal electrostimulation
  Interventions: Other: electrostimulation
- posterior tibial nerve (Experimental): Group treated with transcutaneous electrostimulation of the posterior tibial nerve
  Interventions: Other: electrostimulation
- control (No Intervention): Group of volunteers who will not be treated

INTERVENTIONS:
Other: electrostimulation — Electrostimulation with asymmetric and depolarized biphasic current with a frequency of 10Hz and a pulse width of 200μs.
  Arms: posterior tibial nerve; vaginal

SUMMARY:
This is a clinical trial whose objective is to compare the efficacy of transcutaneous electrostimulation of the posterior tibial nerve with intravaginal electrostimulation in the treatment of women with symptoms of idiopathic overactive bladder. The volunteers will be randomly randomized into three study groups: posterior tibial group, vaginal group and control group. They are evaluated at three times: before the start of treatment, at the end of 6 weeks of treatment and after 1 month (follow up). The evaluation will occur through a voiding diary and a quality of life questionnaire. For the treatment groups will be used depolarized biphasic current with frequency of 10 Hz and pulse width of 200 μs, and intensity according to the tolerance of the patient. The hypothesis of the study is that the two forms of electrostimulation for treatment of idiopathic overactive bladder will be effective, but transcutaneous electrostimulation of the posterior tibial nerve will be more effective than intravaginal.

DETAILED DESCRIPTION:
Objective: To compare the efficacy between intravaginal and transcutaneous electrostimulation of the posterior tibial nerve in the treatment of women with symptoms of idiopathic overactive bladder or mixed urinary incontinence.

METHODS: This is a randomized, controlled, single-blind clinical trial with comparative analysis between study groups and a control, performed at three moments: pre and post clinical intervention and one month after the end of treatment. Vaginal electrostimulation group (GV), transcutaneous electrostimulation group of the posterior tibial nerve (GTP) and control group (CG - without intervention). The intervention groups will be treated with biphasic current with a frequency of 10 Hz and a pulse width of 200 μs for 12 sessions of 30 minutes each. Participants will be evaluated and reevaluated by means of a general data questionnaire, 3-day urinary diary and an International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ-OAB). Statistical analysis will be performed using SPSS version 22 and the level of significance adopted will be p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women
* aged 18 years and over
* literate
* exhibit symptoms of overactive bladder (urinary urgency, urge incontinence, nocturia and polaciuria) or mixed urinary incontinence with predominance of urge incontinence
* to present lower urinary tract dysfunction identified by scores that were equal or higher than 8 points in the Overactive Blader version 8 questionnaire (OAB-V8)
* accept to participate in the study by means of signing the Term of Free and Informed Consent approved by the Research Ethics Committee of the University Hospital of the Northern Region of Paraná State University of Londrina (HURNP / UEL).

Exclusion Criteria:

* Women who are virgin
* pregnant
* have a recurrent lower urinary tract infection (more than three episodes a year)
* vaginal infection
* history of overactive bladder medication in the last three months
* urinary incontinence to efforts exclusively
* previous surgery to treat incontinence urinary
* neurological diseases (such as multiple sclerosis, Alzheimer's disease, stroke, Parkinson's disease)
* current history of genitourinary neoplasia
* genital prolapse above third degree of Baden and Walker
* decompensated diabetic
* patients with cardiac pacemaker
* metal implant in the ankle and right foot
* cognitive deficit that inability to respond to questionnaires properly and / or correctly fill in the voiding diary
* do not perform all treatment sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — age greater than or equal to 18 years
Enrollment: 67 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline miccional emergency at 6 weeks after starting treatment and at 1 month after the end of treatment. | Before starting treatment, 6 weeks after starting treatment and 1 month after the end of treatment.
  Sudden and uncontrollable desire to urinate checked through the voiding diary.

SECONDARY OUTCOMES:
Change from baseline urinary frequency at 6 weeks after starting treatment and at 1 month after the end of treatment. | Before starting treatment, 6 weeks after starting treatment and 1 month after the end of treatment.
  Urinating often (more than 8 events / 24h)
Change from baseline nocturia at 6 weeks after starting treatment and at 1 month after the end of treatment. | Before starting treatment, 6 weeks after starting treatment and 1 month after the end of treatment.
  The necessity wake up 1 or more times during the night to urinate.
Change from baseline urge-incontinence at 6 weeks after starting treatment and at 1 month after the end of treatment. | Before starting treatment, 6 weeks after starting treatment and 1 month after the end of treatment.
  Involuntary loss accompanied or preceded by urine in the immediate aftermath of an emergency episode.
Change from baseline quality of life related to the symptoms of overactive bladder at 6 weeks after starting treatment and at 1 month after the end of treatment. | Before starting treatment, 6 weeks after starting treatment and 1 month after the end of treatment.
  The impact of overactive bladder symptoms on the quality of life of the volunteers will be verified through the International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ-OAB), which is a brief questionnaire with a high psychometric capacity to specifically evaluate overactive bladder. The ICIQ-OAB score ranges from 0 to 16 on a progressive scale, as well as an analog scale from zero to ten to quantify the discomfort caused by each symptom, the higher the score the worse the quality of life.

IPD SHARING:
Plan to Share IPD: No